CLINICAL TRIAL: NCT02850965
Title: Efficacy, Safety, and Immunogenicity of BI 695501 Versus Humira® in Patients With Moderate to Severe Chronic Plaque Psoriasis: A Randomized, Double-Blind, Parallel-Arm, Multiple-Dose, Active Comparator Trial
Brief Title: Efficacy, Safety and Immunogenicity of BI 695501 Versus Humira® in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1297.12; 2016-000613-79 (EudraCT Number)
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — BI 695501; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BI 695501 (Experimental)
  Interventions: Drug: BI 695501
- Humira (Active Comparator)
  Interventions: Drug: Humira

INTERVENTIONS:
Drug: BI 695501
  Arms: BI 695501
Drug: Humira
  Arms: Humira

SUMMARY:
To evaluate the efficacy and to compare efficacy and safety of BI 695501 versus Humira in patients with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Males and females aged >=18 to =<80 years who have a diagnosis of moderate to severe chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study drug (a self-reported diagnosis confirmed by the investigator is acceptable), and which has been stable for the last 2 months with no changes in morphology or significant flares at both Screening and Baseline (Randomization):

  * involved body surface area (BSA) >= 10% and
  * Psoriasis Area and Severity Index (PASI) score >= 12 and
  * static Physician's Global Assessment (sPGA) score of >= 3.
* Participants of reproductive potential (childbearing potential ) must be willing and able to use highly effective methods of birth control per International Council for Harmonization (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly during the trial and for 6 months following completion or discontinuation from the trial medication.
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the trial.
* Patients who are candidates for systemic therapy.

Exclusion criteria:

* Active ongoing inflammatory diseases other than psoriasis that might confound trial evaluations according to investigator's judgment.
* Previous treatment with more than 1 biological agent, or adalimumab or adalimumab biosimilar. No prior biologic exposure within last 6 months of screening.
* Patients with a significant disease other than psoriasis and/or a significant uncontrolled disease (such as, but not limited to, nervous system, renal, hepatic, endocrine, hematological, autoimmune or gastrointestinal disorders).
* Major surgery performed within 12 weeks prior to randomization or planned within 6 months after screening, e.g., total hip replacement.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
* Chronic alcohol or drug abuse
* Women who are pregnant, nursing, or who plan to become pregnant during the course of this study or within the period at least 6 months following completion or discontinuation from the trial.
* Forms of psoriasis (e.g., pustular, erythrodermic and guttate) other than chronic plaque psoriasis. Drug-induced psoriasis (i.e., new onset or current exacerbation from e.g., beta blockers or lithium).
* Primary or secondary immunodeficiency (history of, or currently active), including known history of HIV infection or a positive HIV test at screening (per the investigator discretion and where mandated by local authorities).
* Known chronic or relevant acute tuberculosis; no evidence of active tuberculosis.
* Known clinically significant coronary artery disease, significant cardiac arrhythmias, moderate to severe congestive heart failure (New York Heart Association Classes III or IV) or interstitial lung disease observed on chest X-ray.
* History of a severe allergic reaction, anaphylactic reaction, or hypersensitivity to a previously used biological drug or its excipients.
* Positive serology for hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Receipt of a live/attenuated vaccine within 12 weeks prior to the Screening Visit; patients who are expecting to receive any live/attenuated virus or bacterial vaccinations during the trial or up to 3 months after the last dose of trial drug.
* Any treatment (including biologic therapies) that, in the opinion of the investigator, may place the patient at unacceptable risk during the trial.
* Known active infection of any kind (excluding fungal infections of nail beds), any major episode of infection requiring hospitalization or treatment with intravenous (i.v.) anti infectives within 4 weeks of the Screening Visit
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times upper limit of normal (ULN) at Screening.
* Hemoglobin < 8.0 g/dL at Screening.
* Platelets < 100,000/µL at Screening.
* Leukocyte count < 4000/µL at Screening.
* Creatinine clearance < 60 mL/min/1.73 m2 at Screening.
* Patients with a history of any clinically significant adverse reaction to murine or chimeric proteins, or natural rubber and latex, including serious allergic reactions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (54):
- United States (14):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Alliance Dermatology and MOHS Center PC, Phoenix, Arizona
  - Southern California Dermatology Inc., Santa Ana, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, P.C., Duncansville, Pennsylvania
  - Medical Research South, Charleston, South Carolina
  - Menter Dermatology Research Institute, Dallas, Texas
- Czechia (6):
  - Dorothea, Chomutov
  - MU Dr. Helena Korandova s.r.o., Olomouc-Povel, Olomouc-Povel
  - University Hospital Ostrava, Ostrava
  - HOMEA spol. s.r.o., Pardubice, Pardubice
  - Univ. Hospital Kralovske Vinohrady, Prague
  - MU Dr. Jaroslav Dragon, Ústí nad Labem, Ústí nad Labem
- Estonia (2):
  - Center for Clinical and Basic Research, Tallinn, Tallinn
  - Hospital of South-Estonia Ltd, Võru Maakond, Võru Maakond
- Germany (5):
  - Rothhaar Studien GmbH, Berlin
  - Rosenparkklinik GmbH, Darmstadt, Darmstadt
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Gemeinschaftspraxis Dr. Bräu Dr. Gross, Gießen, Giessen
  - TFS Trial Form Support GmbH, Hamburg
- Poland (11):
  - NZOZ Specderm, Bialystok, Bialystok
  - ClinicMed Badurski i wspolnicy Spolka Jawna, Bialystok, Bialystok
  - NSZOZ Unica CR, Dabrowka, Dąbrówka
  - Synexus Polska SCM Sp. z o.o. Gdansku, Gdansk, Gdansk
  - University Clinical Center, Gdansk, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Gdynia
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Katowice
  - SOLUMED Centrum Medyczne, Poznan, Poznan
  - Laser Clin. S.C. Dr T. Kochanowski Dr A. Krolicki, Szczecin, Szczecin
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warszawa, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Wroclaw
- Russia (8):
  - State Medical University, Kazan, Kazan'
  - LLC Skin Disease Clinic of Pier Volkenstein, St. Petersburg, Saint Petersburg
  - Dermatovenereological Dispensary #10, St. Petersburg, Saint Petersburg
  - ArsVitae NorthWest LLC, Saint Petersburg
  - EKO-Bezopasnost, St. Petersburg, Saint Petersburg
  - 1stPavlov St.Med.Univ.St.-Petersburg Res.Inst., Saint Petersburg
  - Institution of Healthcare "Nikolaevskaya Hospital", Saint Petersburg
  - Smolensk State Medical University, Smolensk, Smolensk
- Slovakia (2):
  - Faculty hospital with clinics F.D. Roosevelta, Banská Bystrica
  - Dermatovenerologicke oddelenie sanatorneho typu, Svidnik, Svidník
- Ukraine (6):
  - Territorial Medical Association Dermatovenerology, Kyiv, Kyiv
  - CH of State Border Service of Ukraine, Lviv, Lviv
  - CI Odesa Regional Dermatovenerologic Dispensary, Odesa, Odesa
  - CI RC Dermatovenerologic Dispensary, Ivano-Frankivsk, Saint Ivano-Frankivsk
  - SI Ternopil Regional Dermatovenerologic Dispensary, Ternopil, Ternopil
  - MCIC MC LLC Health Clinic, Vinnytsia, Vinnytsia

REFERENCES:
- [Derived] Strand V. Summary of Research: Immunogenicity of Adalimumab Reference Product and Adalimumab-adbm in Patients with Rheumatoid Arthritis, Crohn's Disease, and Chronic Plaque Psoriasis: A Pooled Analysis of the VOLTAIRE trials. Rheumatol Ther. 2025 Aug;12(4):613-616. doi: 10.1007/s40744-025-00766-6. Epub 2025 Jun 11. PMID 40498294
- [Derived] Strand V, McCabe D, Bender S. Immunogenicity of adalimumab reference product and adalimumab-adbm in patients with rheumatoid arthritis, Crohn's disease and chronic plaque psoriasis: a pooled analysis of the VOLTAIRE trials. BMJ Open. 2024 Nov 17;14(11):e081687. doi: 10.1136/bmjopen-2023-081687. PMID 39551590
- [Derived] Menter A, Arenberger P, Balser S, Beissert S, Cauthen A, Czeloth N, Soung J, Jazayeri S, Weisenseel P, Jayadeva G. Similar efficacy, safety, and immunogenicity of the biosimilar BI 695501 and adalimumab reference product in patients with moderate-to-severe chronic plaque psoriasis: results from the randomized Phase III VOLTAIRE-PSO study. Expert Opin Biol Ther. 2021 Jan;21(1):87-96. doi: 10.1080/14712598.2021.1851362. Epub 2020 Dec 29. PMID 33317345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase III, multinational, randomized, double-blind, parallel-arm, multiple-dose, active-comparator trial of BI 695501 and US-licensed Humira with a 24-week treatment period and 10 weeks of safety follow up, in patients with moderate to severe chronic plaque psoriasis.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- BI 695501: Patients were administered with BI 695501 via subcutaneous (SC) injection 80 milligram (mg) on Day 1 and 40 milligram (mg) on every other week from Week 1 to Week 23.
- US-licensed Humira: Patients were administered US-licensed Humira via subcutaneous (SC) injection 80 mg on Day 1 and 40 milligram on every other week from Week 1 to Week 23.
Period: Overall Study
Arm/Group | BI 695501 | US-licensed Humira
Started (Randomized) | 159 | 159
Treated | 159 | 158
Completed | 141 | 134
Not Completed | 18 | 25
Not completed — Other than listed | 3 | 4
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 5 | 3
Not completed — Lack of Efficacy | 4 | 8
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): The SAF contained all patients who provided signed informed consent, who were randomized, and who received at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695501 | US-licensed Humira | Total
Number analyzed (Participants) | 159 | 158 | 317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (12.79) | 44.7 (13.92) | 43.4 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 56 | 114
  Male | 101 | 102 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 147 | 146 | 293
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 157 | 156 | 313
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With at Least 75% Reduction in Psoriasis Area and Severity Index (PASI 75) Response at Week 16
Description: The PASI tool provides numeric scoring for a patient's overall psoriasis disease state, ranging from 0 to 72. Head (h), trunk (t), upper extremities (u) and lower extremities (l) areas were assessed; correspond to 10, 30, 20, and 40% of the total body area, respectively. The signs of severity, erythema (E), induration (I) and desquamation (D) of lesions were assessed using a numeric scale of 0 to 4 where 0 was a complete lack of cutaneous involvement and 4 was the severest possible involvement. The area of psoriatic involvement of these areas (Ah, At, Au, and Al) was given a numerical value: 0 = no involvement, 1 = <10%, 2 = 10 to <30%, 3 = 30 to <50%, 4 = 50 to <70%, 5 = 70 to <90%, and 6 = 90 to 100% involvement.
  PASI = 0.1(Eh+Ih+Dh)Ah + 0.3(Et+It+Dt)At + 0.2(Eu+Iu+Du)Au + 0.4(El+Il+Dl)Al.
  Percentage = least squares means per treatment groups back transformed using inverse logit function.
Time Frame: Week 16
Population: Full Analysis Set (FAS): The FAS contained all randomized patients who received at least one dose of trial medication, and had all efficacy measures relevant for the PASI 75, measured at baseline and at least once post-baseline (prior to or on Week 16).
Measure: Number; unit: Percentage (%)
Arm/Group | BI 695501 | US-licensed Humira
Number analyzed (Participants) | 158 | 157
Percentage (%) | 68.2 | 70.4
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira; The week 16 confidence interval for the estimated difference in percentage are produced using the cumulative distribution function method of Reeve; Test type: Equivalence — Protocol defined margins are: [-18.0%, +18.0%] for Week 16, 95% confidence interval. Between-imputation variance is zero. Confidence interval is based on one imputed set; Regression, Logistic; Difference in PASI 75 Response Rate = -2.2, 95% CI 2-sided [-14.4 to 8.7] — Difference in PASI 75 Response Rate = (BI 695501 - US-licensed Humira, %); The statistical model: Logit (response to treatment at Week 16)=Treatment+Baseline PASI+Prior exposure to a biologic agent+random error. Model included fixed, categorical effects of treatment (BI 695501 vs US-licensed Humira) and prior exposure to a biologic agent (yes/no), continuous effect of baseline PASI. The random error was assumed to be binomially distributed

2. Secondary Outcome: The Percentage of Patients With a PASI 75 Response at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: FAS
Measure: Number; unit: Percentage (%)
Arm/Group | BI 695501 | US-licensed Humira
Number analyzed (Participants) | 158 | 157
Percentage (%) | 75.3 | 72.4
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira; The week 24 confidence interval for the estimated difference in percentage are produced using the cumulative distribution function method of Reeve; Test type: Other — Missing PASI 75 at Week 24 data were imputed using a combination of non-responder imputation (NRI) and last observed carried forward (LOCF); Regression, Logistic; Difference in PASI 75 Response Rate = 2.9, 95% CI 2-sided [-8.5 to 12.6] — Difference in PASI 75 Response Rate = (BI 695501 - US-licensed Humira, %); The statistical model: Logit (response to treatment at Week 24)=Treatment+Baseline PASI+Prior exposure to a biologic agent+random error. Model included fixed, categorical effects of treatment (BI 695501 vs US-licensed Humira) and prior exposure to a biologic agent (yes/no), continuous effect of baseline PASI. The random error was assumed to be binomially distributed

3. Secondary Outcome: The Mean Percentage Improvement in PASI at Week 16
Description: The PASI tool provides numeric scoring for a patient's overall psoriasis disease state, ranging from 0 to 72. Head (h), trunk (t), upper extremities (u) and lower extremities (l) areas were assessed; correspond to 10, 30, 20, and 40% of the total body area, respectively. The signs of severity, erythema (E), induration (I) and desquamation (D) of lesions were assessed using a numeric scale of 0 to 4 where 0 was a complete lack of cutaneous involvement and 4 was the severest possible involvement. The area of psoriatic involvement of these areas (Ah, At, Au, and Al) was given a numerical value: 0 = no involvement, 1 =<10%, 2 =10 to <30%, 3 =30 to <50%, 4 =50 to <70%, 5 =70 to <90%, and 6 =90 to 100% involvement.
  PASI = 0.1(Eh+Ih+Dh)Ah + 0.3(Et+It+Dt)At + 0.2(Eu+Iu+Du)Au + 0.4(El+Il+Dl)Al.
  Results based on PASI mean percentage improvement from Baseline after 16 weeks of treatment = overall mean + treatment group + Baseline PASI + prior exposure to a biological agent + random error.
Time Frame: Week 16
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage (%)
Arm/Group | BI 695501 | US-licensed Humira
Number analyzed (Participants) | 149 | 149
Percentage (%) | 83.7 [80.2 to 87.2] | 82.1 [78.6 to 85.6]
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira; Analysis of covariance (ANCOVA) was performed based on the following model: PASI percentage improvement from baseline at Week 16= Treatment + Baseline PASI +Prior exposure to a biologic agent + random error; Test type: Other; ANCOVA; Analysis of covariance (ANCOVA); Difference of Least Squares Means = 1.7, 95% CI 2-sided [-2.7 to 6.0] — Difference of Least Squares Means (LSM)= LSM of (BI 695501 - Humira)

4. Secondary Outcome: The Percentage of Patients With a Static Physician's Global Assessment (sPGA) ≤1 (Clear or Almost Clear) at Week 16
Description: The Static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions.
  The assessment was considered "static", which referred to the patient's disease state at the time of the assessment, without comparison to any of the patient's previous disease states (dynamic), whether at Baseline or at a previous visit. A lower score indicated less body coverage, with 0 being clear, 1 being almost clear, and 4 being.
  Percentage = least squares means per treatment groups back transformed using inverse logit function.
Time Frame: Week 16
Population: FAS
Measure: Number; unit: Percentage (%)
Arm/Group | BI 695501 | US-licensed Humira
Number analyzed (Participants) | 158 | 157
Percentage (%) | 59.6 | 52.1
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira; [analysis description as in outcome 1, analysis 1]; Test type: Other — Missing sPGA at Week 16 data were imputed using a combination of non-responder imputation (NRI) and last observed carried forward (LOCF); Regression, Logistic; Difference in sPGA <= 1 Response Rate = 7.5, 95% CI 2-sided [-4.8 to 19.1] — Difference in sPGA <= 1 Response Rate = (BI 695501 - US-licensed Humira, %); The statistical model: Logit (response to treatment at Week 16)=Treatment+Baseline PASI+Prior exposure to a biologic agent+random error. Model included fixed, categorical effects of treatment (BI 695501 vs US-licensed Humira) and prior exposure to a biologic agent (yes/no), continuous effect of baseline PASI

5. Secondary Outcome: The Percentage of Patients Achieving a Dermatology Life Quality Index (DLQI) of 0 or 1 at Week 16
Description: The DLQI is a subject-administered, 10-question, that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. It has a 1-week recall period. Every item score ranges from 0 (not relevant/not at all) to 3 (very much). Question 7 is a "yes/no" question where "yes" is scored as 3.
  The DLQI total score was calculated by summing the scores of each question resulting in a range of 0 to 30 where 0-1 = no effect on subject's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on the subject's life.
  The higher the score, the more the quality of life is impaired. If the answer to 1 question in a domain was missing, that domain was treated as missing. If 2 or more questions were left unanswered (missing), DLQI total score was treated as missing. Percentage = least squares means per treatment groups back transformed using inverse logit function.
Time Frame: Week 16
Population: FAS
Measure: Number; unit: Percentage (%)
Arm/Group | BI 695501 | US-licensed Humira
Number analyzed (Participants) | 158 | 157
Percentage (%) | 67.2 | 66.8
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira; [analysis description as in outcome 1, analysis 1]; Test type: Other — Missing DLQI at Week 16 data were imputed using a combination of non-responder imputation (NRI) and last observed carried forward (LOCF); Regression, Logistic; Difference in DLQI Response Rate = 0.4, 95% CI 2-sided [-11.7 to 11.3] — Difference in DLQI (0, 1) Response Rate = (BI 695501 - US-licensed Humira, %); [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: The Percentage of Patients With Drug-related Adverse Events (AEs)
Description: The secondary safety endpoint was defined as the percentage of patients with drug-related adverse events (AEs).
Time Frame: From first drug administration until 10 weeks after last drug administration, up to 34 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients (%)
Arm/Group | BI 695501 | US-licensed Humira
Number analyzed (Participants) | 159 | 158
Percentage of patients (%) | 13.2 | 20.3

ADVERSE EVENTS:
Time Frame: From first drug administration until 10 weeks after last drug administration, up to 33 weeks.
Arm/Group | BI 695501 | US-licensed Humira
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/158
Serious Adverse Events (participants affected / at risk) | 5/159 | 7/158
Other Adverse Events (participants affected / at risk) | 17/159 | 24/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (N=159) | US-licensed Humira (N=158)
Abdominal abscess (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (N=159) | US-licensed Humira (N=158)
Nasopharyngitis (Infections and infestations) | 12 | 7
Injection site erythema (General disorders) | 5 | 10
Injection site pain (General disorders) | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT02850965/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT02850965/SAP_001.pdf